CLINICAL TRIAL: NCT03767075
Title: Basket of Baskets: A Modular, Open-label, Phase II, Multicentre Study To Evaluate Targeted Agents in Molecularly Selected Populations With Advanced Solid Tumours
Brief Title: A Modular Multi-Basket Trial to Improve Personalized Medicine in Cancer Patients (Basket of Baskets)
Acronym: BoB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Collaborators: Roche Pharma AG (Industry); Iqvia Pty Ltd (Industry); Taisho Pharmaceutical Co., Ltd. (Industry); Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHIO17002; 2017-005108-89 (EudraCT Number)
Record Dates: First submitted 2018-11-14; First posted 2018-12-06 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor; Cancer; Atezolizumab; Immunotherapy
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; futibatinib; amivantamab

STUDY DESIGN:
Intervention Model Description: * Part A includes a molecular profiling program for subjects with advanced solid tumors (iPROFILER) and a molecular tumor board to select the most appropriate treatment based on the molecular alterations found in the iPROFILER.
  * Part B includes iBASKET, a modular investigator initiated basket study for subjects with selected molecular alterations.
Masking Description: no masking is used. All involved know the identity of the intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Module 1 - Atezolizumab (Experimental): Genomically selected populations will all receive the same drug
  * Arm 1A: BRCA1 or BRCA2 mutations
  * Arm 1B: MLH1, MSH2, MSH6, or PMS2 mutations
  * Arm 1C: tumors with POLE mutation, POLD1 mutation
  * Arm 1D: hypermutated tumors
  * Arm 1E: tumors with other mutations in DNA-repair genes
  * Arm 1F: tumors with amplified PDL1
  * Arm 1G: tumours with CDK12 mutations
  Subjects will be recruited and allocated to arms according to their biomarker profile. It is assumed that 1000 subjects will need to be screened in part A in order to enroll 120 patients in part B of module 1.
  Interventions: Drug: Atezolizumab
- Module 2 - Futibatinib (Experimental): Genomically selected populations will all receive the same drug
  * Arm 2A: Known pathogenic FGFR1-3 mutations
  * Arm 2B: Variants of unknown significance in FGFR1-3 with functional relevance or pathogenic FGFR4 mutations.
  * Arm 2C: Highly amplified FGFR1-3 with high FGFR1-3 mRNA (with the exception of gastric and breast cancer)
  * Arm 2D: Highly amplifiedFGFR1-3 without high FGFR1-3 mRNA (with the exception of gastric and breast cancer)
  Subjects will be recruited and allocated to arms according to their biomarker profile. It is assumed that 2000 subjects will need to be screened in part A in order to enroll 80 patients in part B of module 2.
  Interventions: Drug: Futibatinib
- Module 3 - Amivantamab (Experimental): Genomically selected populations will all receive the same drug
  * Arm 3A: kinase domain mutations/ MET fusion-genes (including intragene exon skipping MET-MET fusions)
  * Arm 3B: MET copy number gain (equivalent CNG ≥6) (exception: colorectal cancer)
  * Arm 3C: EGFR mutations (exception: primary lung malignancies)
  Subjects will be recruited and allocated to arms according to their biomarker profile. It is assumed that 1725 subjects will need to be screened in part A in order to enroll 69 patients in part B of module 3.
  Interventions: Drug: Amivantamab

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg, administered IV, once every 3 weeks
  Arms: Module 1 - Atezolizumab
Drug: Futibatinib — 20 mg administered orally, once daily (QD) continuously in 28-day cycles.
  Other Names: TAS-120
  Arms: Module 2 - Futibatinib
Drug: Amivantamab — 1050 mg administered IV for body weight < 80 kg and 1400 mg for body weight >= 80 kg mg once weekly in Cycle 1 (with a split dose on Days 1-2) and then every 2 weeks in subsequent cycles (28-day cycles)
  Other Names: JNJ-372
  Arms: Module 3 - Amivantamab

SUMMARY:
The global objective of this Basket of Basket study is to evaluate the antitumor activity of each matched therapies that will be evaluated through the study in small molecularly selected populations.

The objective of module 1 wil be to determine the overall response rate (ORR) at 12 weeks by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of atezolizumab in each of the arms of the module. All patients in genomically selected populations will receive atezolizumab 1200 mg IV every 3 weeks.

The objective of module 2 wil be to determine the overall response rate (ORR) at 16 weeks by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of futibatinib in each of the arms of the module. All patients in genomically selected populations will receive will receive futibatinib, 20 mg, once daily (QD) in 28-day cycles.

The objective of module 3 wil be to determine the overall response rate (ORR) at 12 weeks by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of amivantamab in each of the arms of the module. All patients in genomically selected populations will receive amivantamab 1050 mg intravenously (IV) for body weight < 80 kg and 1400 mg for body weight >= 80 kg mg once weekly in Cycle 1 (with a split dose on Days 1-2) and then every 2 weeks in subsequent cycles (28-day cycles).

DETAILED DESCRIPTION:
Basket studies are a new sort of clinical studies to identify patients with the same kind of mutations and treat them with the same drug, irrespective of their specific cancer type. In basket studies, depending on the mutation types, patients are classified into "baskets". Targeted therapies that block that mutation are then identified and assigned to baskets where patients are treated accordingly.

This protocol has two parts: part A (iPROFILER), which includes the common procedures for tumor molecular profiling and treatment recommendation, and part B (iBASKET), which corresponds to the therapeutic portion.

The purpose of part A (iPROFILER) of this study is to test participants' tumour tissue in order to identify whether their tumour has certain mutations in cancer-related genes. It is known that gene mutations of tumours contribute to their origin and growth and determine whether the tumour will respond to particular cancer drugs. This test will provide information about potential targeted therapies that specifically attack those gene mutations. The purpose of part B (iBASKET) of this study is to offer participants a personalised anti-cancer treatment based on the gene mutations that are found in their tumour.

Participants taking part in module 1 of part B (iBASKET) will receive atezolizumab 1200 mg IV every 3 weeks, following the analysis of their tumour in part A (iPROFILER). Participants will be able to take atezolizumab for as long as their tumour doesn't grow and for as long as they don't have any side-effects which prevent them from continuing treatment. Module 1 will have a 2-year recruitment period. The aim of the study is to determine which genomically selected populations respond effectively to the targeted treatment, atezolizumab. Approximately 1000 participants will be enrolled into part A (iPROFILER), with approximately 120 participants being recruited into module 1 of part B (iBASKET).

Participants taking part in module 2 of part B (iBASKET) will receive will receive futibatinib, 20 mg, once daily (QD) in 28-day cycles, following the analysis of their tumour in part A (iPROFILER). Participants will be able to take futibatinib for as long as their tumour doesn't grow and for as long as they don't have any side-effects which prevent them from continuing treatment. Module 2 will have a 2-year recruitment period. The aim of the study is to determine which genomically selected populations respond effectively to the targeted treatment, futibatinib. Approximately 1000 participants will be enrolled into part A (iPROFILER), with approximately 80 participants being recruited into module 2 of part B (iBASKET).

Participants taking part in module 3 of part B (iBASKET) will receive amivantamab 1050 mg IV for body weight < 80 kg and 1400 mg for body weight >= 80 kg mg once weekly in Cycle 1 (with a split dose on Days 1-2) and then every 2 weeks in subsequent cycles (28-day cycles), following the analysis of their tumour in part A (iPROFILER). Participants will be able to take amivantamab for as long as their tumour doesn't grow and for as long as they don't have any side-effects which prevent them from continuing treatment. Module 3 will have a 2.5-year recruitment period. The aim of the study is to determine which genomically selected populations respond effectively to the targeted treatment, amivantamab. Approximately 1725 participants will be enrolled into part A (iPROFILER), with approximately 69 participants being recruited into module 3 of part B (iBASKET).

ELIGIBILITY:
Eligibilty Criteria (PART A - iPROFILER)

Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed malignancy that is metastatic or unresectable, who have progressed to standard therapy, who are receiving a standard anticancer treatment, but no subsequent approved treatment would be available upon progression, who are unable to receive standard therapy, or for whom standard therapy does not exist.
2. Patient must have ECOG performance status of 0 or 1.
3. Subjects must be 18-year-old or older.
4. Subjects must have measurable disease according to RECIST 1.1.
5. Subjects must have enough tumour tissue for molecular analysis.

   1. Subjects providing formalin-fixed paraffin embedded tissue (FFPE) must provide a minimum amount of tissue ranging from 28 to 36 slides depending on the sample tumour cellularity. If there is not enough archival tissue to meet this criterion, the patient must undergo a tumour biopsy.
   2. Subjects providing fresh frozen tissue must provide 5 core biopsies or equivalent.

      Fresh frozen tissue must be preferentially collected from a tumour biopsy; hence, subjects must have disease amenable to be biopsied. Otherwise, the patient should have fresh frozen tumour tissue stored in a biobank or biorepository.
   3. Efforts will be made to provide fresh frozen tissue in at least one quarter of the participating subjects. The proportion of subjects that might provide fresh frozen tissue might change based on the results from the molecular analysis.
   4. Since some of the tests are performed in FFPE tissue, subjects providing fresh frozen tissue from a recent biopsy will have part of the sample processed in FFPE as per Laboratory manual.
6. Subjects must have adequate haematological, renal, and hepatic function.
7. For subjects requiring a tumour biopsy: subjects must have adequate coagulation function.
8. Subjects must be willing to participate in a clinical trial with a matched therapy according to the molecular profile of his/her tumour.

Exclusion Criteria:

1. Subjects with leptomeningeal disease should be excluded from this clinical trial.
2. Subjects with known unstable brain metastases should be excluded from this clinical trial. Exception: Subjects who have undergone surgery and/or radiotherapy and in which brain metastases remain stable or decrease in size for six months after having completed therapy.
3. Subjects with spinal cord compression not definitively treated with surgery and/or radiation.
4. Subjects with uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure, LVEF < 50%, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Subjects with inability to swallow tablets or capsules.
6. Subjects with known HIV, hepatitis B or hepatitis C infection.
7. Subjects with known history of malabsorption.

Eligibilty Criteria (PART B - iBASKET)

Inclusion Criteria:

1. Subjects must have metastatic or unresectable malignant tumour, histologically or cytological confirmed and progressing to current therapy. Tumours must be refractory to standard therapy or for which standard therapy does not exist, or subjects may be unable to receive standard therapy.
2. Patient must have ECOG performance status of 0 or 1.
3. Subjects must be 18-year-old or older.
4. Subjects must have measurable disease according to RECIST 1.1.
5. Subjects must be willing to participate in a clinical trial with a matched therapy according to the molecular profile of his/her tumour.
6. Tumours must harbour the following alterations.
7. Subjects must have adequate hematological, renal, and hepatic function.
8. For subjects requiring a tumour biopsy: subjects must have adequate coagulation function.
9. A woman of childbearing potential must have a negative serum pregnancy test within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy test during the study.
10. A woman must be either of the following:

    1. Not of childbearing potential.
    2. Of childbearing potential and practicing true abstinence during the entire period of the study, including up to 6 months after the last dose of study treatment is given.
    3. Of childbearing potential and practicing 2 methods of contraception, including 1 highly effective user independent method and a second method. Participant must agree to continue contraception throughout the study and through 6 months after the last dose of study treatment.
11. A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study treatment.
12. A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 6 months after receiving the last dose of study treatment.
13. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Pregnant or breastfeeding women. Females of childbearing potential must have a negative serum pregnancy test within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy test during the study.
2. Any approved anticancer therapy, including chemotherapy, hormonal therapy or radiotherapy, within 3 weeks prior to initiation of study treatment; however, the following are allowed:

   1. Hormone-replacement therapy or oral contraceptives.
   2. Somatostatin analogues for the treatment of symptoms related with neuroendocrine tumours.
   3. Gonadotropin-releasing hormone agonists or antiandrogens for prostate cancer.
   4. Palliative radiotherapy for bone metastases > 2 weeks prior to Cycle 1, Day 1.
3. Treatment with an investigational agent within 3 weeks prior to Cycle 1, Day 1 (or within five half-lives of the investigational product, whichever is longer).
4. Patients with recent major surgery or invasive procedure within 15 days before the fist dose of the study drug.
5. Participant has unstable symptomatic brain metastases. A participant with asymptomatic or previously treated and stable brain metastases may participate in this study.

   a. Participants who have received definitive radiation or surgical treatment for symptomatic or unstable brain metastases and have been clinically stable and asymptomatic for at least 2 weeks before enrolment are eligible, provided they have been either off corticosteroid treatment or are stable or tapering doses below 4 mg of dexamethasone.
6. Patients with meningeal or leptomeningeal carcinomatosis.
7. Uncontrolled intercurrent illness including, but not limited to, active infection, cardiovascular disease, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg). Note: Subjects with a prior history of HBV demonstrated by positive hepatitis B core antibody are eligible if they have at Screening 1) a negative HBsAg and 2) an HBV DNA (viral load) below the lower limit of quantification, per local testing.
9. Positive hepatitis C antibody (anti-HCV). Note: Subjects with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.
10. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class III or greater), myocardial infarction within 3 months prior to Cycle 1, Day 1, unstable angina or unstable clinically meaningful arrhythmias.
11. Another primary malignancy other than disease under study within 2 years prior to Cycle 1 Day 1, unless consider at low risk of relapse at Investigator discretion.
12. Contraindications included in the product information of the drugs used in the study.

Other protocol specified criteria for each module. The study center will determine if criteria for participation are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | From the first dose date of study treatment to first CR or PR, whichever came earlier, up to 12 weeks (Module 1 & 3) and 16 weeks (Module 2)
  Proportion of patients with a partial response [PR] or complete response [CR] per RECIST v1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS by RECIST 1.1) | From initiation of treatment to objective progression or death from any cause, whichever occurs first, up to two years
  Time from the first dose date of study treatment to the date of investigator-determined objective progression (according to RECIST 1.1) or death from any cause, whichever occurs first.
Overall Survival | From initiation of treatment to death from any cause, up to two years
  Time from beginning treatment to the time of death from any cause.
Duration of response | From documentation of the first CR or PR to the time of first documented evidence of progressive disease (or relapse for subjects who experience CR during the study) or death (up to apprixmatelly 6 months).
  Time from documentation of the first CR or PR to the time of first documented evidence of progressive disease (or relapse for subjects who experience CR during the study) or death.
Health-related quality of life (HRQoL) | Baseline up to data cut-off, up to two years.
  Assessed with the European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30)
Incidence and severity of adverse events | From initiation of treatment to 30 days (all adverse events), and 90 days (all SAEs and AESIs), then any SAE considered treatment-related.
  Type, incidence, severity, timing, seriousness, and relatedness of adverse events and laboratory abnormalities, graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Rodon, MD, Study Chair — MD Anderson
Locations (8):
- Institut Gustave Roussy, Villejuif, France
- Germany (2):
  - Deutsches Krebsforschungszentrum (NCT/DKFZ), Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Dresden, Dresden
- Instituto Nazionale dei Tumori di Milano, Milan, Italy
- Nederland Kanker Instituut (NKI), Amsterdam, Netherlands
- Hospital Vall d'Hebron, Barcelona, Spain
- Karolinska University Hospital Solna, Stockholm, Sweden
- Cancer Research UK Cambridge Centre, Cambridge, United Kingdom